CLINICAL TRIAL: NCT04956211
Title: Systemic Effects of Periodontal Therapy on Patients With Ischemic Stroke. A Pilot Randomized Controlled Clinical Trial
Brief Title: Periodontal Treatment and Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Yago Leira Feijoo, Principal Investigator, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP1
Record Dates: First submitted 2021-06-15; First posted 2021-07-09 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Stroke, Ischemic; Periodontitis
Keywords: endothelium; inflammation; recurrence
MeSH Terms: conditions — Ischemic Stroke; Periodontitis; Inflammation; Recurrence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-surgical periodontal therapy (Experimental): Oral hygiene instructions will be given to all individuals. Any hopeless tooth or categorised as irrational to treat at baseline visit will be extracted at the treatment visit(s). Patients will receive a standard regimen of scaling and root planing of the root surfaces under local analgesia (depending on the severity in one or two sessions within 2 days) with curettes and ultrasonic instruments .
  Interventions: Procedure: Periodontal therapy
- Conventional periodontal therapy (Active Comparator): Oral hygiene instructions will be given to all individuals. Any hopeless tooth or categorised as irrational to treat at baseline visit will be extracted at the treatment visit(s). Supragingival cleaning and polishing of all dentition will be delivered to individuals in this group.
  Interventions: Procedure: Periodontal therapy

INTERVENTIONS:
Procedure: Periodontal therapy — Patients will receive a standard regimen of scaling and root planing of the root surfaces under local analgesia (depending on the severity in one or two sessions within 2 days) with curettes and ultrasonic instruments.

SUMMARY:
A bulk of observational evidence suggests an association between periodontitis and recurrent vascular events in ischemic stroke survivors. One plausible biological mechanism relies on the systemic inflammatory response posed by periodontitis together with changes in the normal function of the vascular endothelium which might lead to recurrence in these population. A non-pharmacological anti-inflammatory treatment (non-surgical periodontal therapy) has shown to reduce systemic inflammatory markers and improve endothelial function. Therefore, we propose to carry out a 1-year follow-up pilot randomized controlled clinical trial to investigate whether control of local and systemic inflammation as well as improve function of the vascular endothelium can lead to reduce the risk of recurrence in patients diagnosed from ischemic stroke.

DETAILED DESCRIPTION:
Every year 71,780 Spaniards develop an stroke and of these 13% do not survive, which makes this disease the second most common cause of death in Spain. Within stroke survivors, it is estimated that 30% are left with some type of disability. The most common type of stroke is ischemic (corresponding to 80% of total stroke cases) which is caused by obstruction of cerebral arteries or by a clot that forms within the brain's own blood vessel or by a clot that is produced elsewhere in the circulatory system and travels to the brain. One of the main factors that contribute to increased morbidity and mortality and hospitalization in stroke patients are recurrent vascular events (RVE) (ie acute myocardial infarction, new stroke / transient ischemic attack or death due to vascular causes). Depending on the stroke subtype, study population and study follow-up, RVEs occur between 1% and 25%. Therefore, the prevention and/or reduction of the number of RVE after stroke would significantly reduce the large accumulated public health burden associated with this type of neurological disease.

The systemic inflammatory response plays a key role in focal cerebral ischemia and in the mechanisms of progression of cerebral infarction, as it is associated with an increased risk of stroke and RVE after a first ischemic stroke. In fact, markers of systemic inflammation such as interleukin 6 (IL-6), C-reactive protein (CRP) or tumor necrosis factor alpha (TNF-α) have been shown to be stroke predictors capable of modifying stroke risk by themselves as well as the risk of suffering a stroke regardless of conventional vascular risk factors. On the other hand, atherosclerosis is considered today as an inflammatory disease and contributes to a large proportion of strokes, both directly due to large vessel atherosclerosis and indirectly due to cardioembolism as a result of cardiac arrhythmias caused by coronary artery disease or emboli after myocardial infarction. A prospective cohort study demonstrated that elevated levels of IL-6 in peripheral blood is a good predictor of future RVE in stroke patients. In addition, one of the links between potential vascular risk factors, systemic inflammation, platelet activation, atherosclerosis and subsequently the appearance of cerebral infarcts is endothelial dysfunction characterized by a reduction in the biological capacity of the endothelium. In this sense, endothelial dysfunction measured by flow-mediated vasodilation (FMD) in the brachial artery is considered a predictor of future vascular complications.

Periodontitis is an immuno-inflammatory disease caused by oral bacteria that is characterized by the destruction of the supporting tissues of the tooth (gum and bone) that, if left untreated, can lead to tooth loss. In Spain, it is estimated that only 5% of the adult population has healthy gums, more than half suffer from gingivitis (reversible inflammation of the gingiva) and an average 38% have periodontitis, increasing this figure to 65% in the elderly 55 years. Worldwide, the most advanced forms of the disease are considered the sixth most prevalent disease in humans, affecting approximately 11% of the adult population worldwide. The main problem with periodontitis is that the harmful effects that produces are not only confined to the oral cavity but also have systemic effects. A meta-analysis of epidemiological studies has found that patients with advanced periodontitis have almost 3-fold increased risk of having large vessel ischemic stroke compared to those without periodontitis. Similar data have been obtained for cerebral small vessel disease (ie, lacunar infarction). Furthermore, in patients who have already had an ischemic stroke, the risk of suffering a second vascular event after two years of follow-up is 2 times higher in those with advanced periodontitis compared to subjects with healthy gums.

Non-surgical periodontal treatment has proven to be a safe and effective non-pharmacological treatment model for not only controlling periodontal infection and inflammation, but is also capable of reducing inflammation at the systemic level (peripheral levels of IL-6 and CRP) as well as improving endothelial function (measured by FMD).

Due to the fact that there is a solid epidemiological relationship between both pathologies and that an increase in the systemic inflammatory response and endothelial dysfunction may be possible mechanisms involved in this association, as well as in the increased risk of RVE development in this population, we propose to carry out a pilot randomized controlled clinical trial to evaluate the effect of non-surgical periodontal treatment on markers of systemic inflammation, endothelial function as well as stroke recurrence in patients with ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years old.
* Non-severely disabling initial ischemic stroke (mRS≤3) in the last 90 days.
* With diagnosis of severe periodontitis (generalized stage III-IV).
* Presence of at least 10 teeth in the mouth.

Exclusion Criteria:

* Patients receiving periodontal treatment in the last 12 months.
* Stroke due to intracranial hemorrhage, dissection, veno-occlusive disease, drugs, trauma or vasculitis.
* Previous neurological impairment that would make detection of a subsequent event difficult.
* Comorbidities that may limit survival <12 months.
* Brain CT/MRI that shows a lesion other than stroke as a cause of syndrome.
* History of medical conditions requiring antibiotic prophylaxis prior to dental exam.
* Pregnants or breastfeeding.
* Known allergy or hypersensitivity to local anesthesia thst cannot be medically managed.
* Patients with bleeding disorders or

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-11-11 (Estimated); Study Completion 2023-12-29 (Estimated)

PRIMARY OUTCOMES:
IL-6 serum levels | from baseline to 6 months after therapy
  Concentrations of IL-6 in serum will be measured by ELISA technique

SECONDARY OUTCOMES:
Other inflammatory markers | from baseline to 6 months after therapy
  Concentrations of hs-CRP, TNF-alpha and IL-1beta in serum will be measured by ELISA technique
Flow-mediated dilatation (brachial artery) | from baseline to 6 months after therapy
  After detection of brachial artery vasomotion, ultrasound evaluation will be made on the dominant forearm. Two-dimensional brachial artery imaging and measurements were performed in all patients by the same operator. Straight segments of the artery will be chosen above the antecubital fosse, perpendicular to the ultrasound beam and along its long axis. Flow-mediated dilatation caused by shear-induced endothelial nitric oxide production will be detected after occlusion of the forearm circulation. A longitudinal image will be used to measure brachial artery diameter; a blood pressure cuff will be inflated on the upper arm to 300 mmHg for 4 min and then deflated, and after 45 s to 1 min, a second longitudinal scan will be obtained, to calculate the brachial artery diameter.
Intima-media thickness (carotid artery) | from baseline to 6 months after therapy
  The image will be focused on the posterior (far) wall of the left carotid artery. A minimum of four measurements of the common carotid far wall was taken 10 mm proximal to the bifurcation, to derive the mean carotid intima-media thickness. The presence of an atheroma plaque will be evaluated in the common and internal carotid extracranial arteries as well as the bifurcations according to standardized scanning and reading protocols. Plaque will be defined as a focal structure that encroaches into the arterial lumen at least 0.5 mm or 50% of the surrounding intima-media thickness value, or demonstrates a thickness >1.5 mm as measured from the media-adventitia interface to the intima-lumen interface.
Recurrent vascular events | from baseline to 12 months after therapy
  Recurrent vascular events will be defined as the development of recurrent stroke, coronary events, peripheral arterial disease, and cardiovascular death during the study period in the present study. Recurrent stroke will be defined as the development of a new focal neurologic deficit or new deterioration of a previous deficit accompanied by a de novo imaging evidence of brain infarction, but the development of transient ischemic attack or hemorrhagic transformation of the previous infarct lesion will be excluded in our present study. Coronary event will be defined as the development of obstructive atherosclerotic coronary artery disease (% diameter stenosis >70%) or myocardial infarction demonstrated by conventional coronary or cardiac CT angiography. Peripheral arterial disease is defined as the development of a narrowing of the arteries other than those that supply the heart or the brain with an ankle brachial index <0.9.
Lipid fractions | from baseline to 6 months after therapy
  Total cholesterol, HDL, LDL and triglycerides will be measured in serum.
Blood pressure | from baseline to 12 months after therapy
  Systolic and diastolic blood pressure measurement will be recorded following recent clinical guidelines using an automated device.
Metabolic control I | from baseline to 6 months after therapy
  HbA1c will be recorded following recent clinical guidelines using an automated device.
Metabolic control II | from baseline to 6 months after therapy
  Blood glucose will be measured in serum

CONTACTS AND LOCATIONS:
Overall Officials: Yago Leira, PhD, Principal Investigator — Health Research Institute of Santiago
Locations (1):
- University of Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ye Z, Cao Y, Miao C, Liu W, Dong L, Lv Z, Iheozor-Ejiofor Z, Li C. Periodontal therapy for primary or secondary prevention of cardiovascular disease in people with periodontitis. Cochrane Database Syst Rev. 2022 Oct 4;10(10):CD009197. doi: 10.1002/14651858.CD009197.pub5. PMID 36194420